CLINICAL TRIAL: NCT02292030
Title: Cardioversion of Atrial Fibrillation Accompanied by Chronic Heart Faliure With or Without HTEA
Brief Title: Cardioversion of Atrial Fibrillation Accompanied by Chronic Heart Faliure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Wei Liu, Prof., Harbin Medical University
Other Study IDs: dong hao
Record Dates: First submitted 2014-11-09; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cardioversion+HTEA: Heart failure patients accompanied by atrial fibrillation receive the treatment of cardioversion+HTEA.
  Interventions: Drug: HTEA
- only cardioversion: Heart failure patients accompanied by atrial fibrillation receive the treatment of cardioversion, but not with HTEA.
  Interventions: Drug: HTEA

INTERVENTIONS:
Drug: HTEA — usually high thoracic epidural anesthesia
  Other Names: High thoracic epidural anesthesia

SUMMARY:
The purpose of this study is to explore the efficacy of low energy cardioversion on atrial fibrillation accompanied with chronic heart failure treated with HTEA or usual medicine.

DETAILED DESCRIPTION:
The purpose of this study is to explore the efficacy of low energy (30J) cardioversion on atrial fibrillation accompanied with chronic heart failure treated with HTEA or usual medicine.

ELIGIBILITY:
Inclusion Criteria:

* congestive heart failure accompanied by atrial fibrillation.

Exclusion Criteria:

* Valvular heart diseases.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: congestive heart failure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
recurrence of atrial fibrillation | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ren Xiaohui, Harbin, Heilongjiang
  - the first affiliated hospital of Harbin Medical University, Harbin, Heilongjiang